CLINICAL TRIAL: NCT00842543
Title: Effects Of A Fruit And Vegetable Juice Concentrate (FVJC) In-Vivo On Retinol Binding Protein 4 And Antioxidant Capacity In Normal And Overweight Boys -A Pilot Randomized Placebo Controlled Study
Brief Title: Fruit and Vegetable Juice Concentrate Effects on RBP4 and Antioxidant Capacity in Lean and Overweight 6-10 Year Old Boys
Acronym: FVJC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: NSA, LLC (Industry)
Responsible Party: Principal Investigator, Jose Atilio Canas, MD, Principal Investigator, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1607330001
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Obesity
Keywords: Nutrition; Oxidative Stress; Insulin Resistance; Whole Food Supplement; Pediatric; Retinoids; Antioxidants; Dietary Supplements
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Fruit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Overweight (Experimental): Overweight Boys receiving either Fruit and Vegetable Juice Concentrate (FVJC) or Placebo, 1 capsule, twice a day, for 6 months
  Interventions: Dietary Supplement: Fruit and Vegetable Juice Concentrate (FVJC); Dietary Supplement: Placebo
- Lean (Experimental): Lean Boys receiving either Fruit and Vegetable Juice Concentrate (FVJC) or Placebo, 1 capsule, twice a day, for 6 months
  Interventions: Dietary Supplement: Fruit and Vegetable Juice Concentrate (FVJC); Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fruit and Vegetable Juice Concentrate (FVJC) — Take FVJC or placebo twice a day for 6 months while receiving dietary and physical activity counseling from a Registered Dietician.
Dietary Supplement: Placebo — Take FVJC or placebo twice a day for 6 months while receiving dietary and physical activity counseling from a Registered Dietician.

SUMMARY:
Our study aims to evaluate if the consumption of a Fruit and Vegetable Juice Concentrate (FVJC) vs. placebo can exert changes in the serum levels of Retinol Binding Protein 4 (RBP4), carotenoids, tocopherol, antioxidant capacity, pro-inflammatory markers, insulin sensitivity in conjunction with weight management in a cohort of lean as compared to overweight healthy six to ten year-old boys. The boys will undergo a detailed medical and family history and a complete physical examination during the screening visit. Careful anthropometric measures and body composition by DEXA will be performed. Nutritional and exercise counseling will be given at the start of the study. The outcome measures will include differences in serum RBP4, antioxidant levels, inflammatory markers and insulin sensitivity at baseline and six months after consumption of FVJC in a randomized double blind placebo control manner.

ELIGIBILITY:
Inclusion Criteria:

* 6-10 year old healthy boys
* Lean or overweight
* Have not started puberty

Exclusion Criteria:

* Chronic illness, asthma, or GI disorder
* Vegan Diet
* Use of routine medications or vitamins 4 weeks before study

Ages: 6 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atilio Canas, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Result] Canas JA, Damaso L, Altomare A, Killen K, Hossain J, Balagopal PB. Insulin resistance and adiposity in relation to serum beta-carotene levels. J Pediatr. 2012 Jul;161(1):58-64.e1-2. doi: 10.1016/j.jpeds.2012.01.030. Epub 2012 Feb 28. PMID 22381025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from pediatric endocrinology clinics, in Jacksonville, USA between July 2008 and December 2009.
Pre-assignment Details: Of the 246 children screened for eligibility, 74 did not meet criteria, 35 refused to participate, 98 were not randomized for various reasons, 39 were randomized.
Groups:
- Overweight FVJC: Overweight Boys prior to receiving Fruit and Vegetable Juice Concentrate (FVJC), 1 capsule, twice a day, for 6 months.
- Lean FVJC: Lean Boys prior to receiving Fruit and Vegetable Juice Concentrate (FVJC), 1 capsule, twice a day, for 6 months.
- Overweight Placebo; Lean Placebo: Lean Boys prior to receiving Placebo, 1 capsule, twice a day, for 6 months.
Period: Overall Study
Arm/Group | Overweight FVJC | Lean FVJC | Overweight Placebo | Lean Placebo
Started | 13 | 5 | 13 | 8
Completed | 11 | 5 | 10 | 4
Not Completed | 2 | 0 | 3 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Overweight Placebo: Overweight Boys prior to receiving Placebo, 1 capsule, twice a day, for 6 months.
- Total: Total of all reporting groups
Arm/Group | Overweight FVJC | Lean FVJC | Overweight Placebo | Lean Placebo | Total
Number analyzed (Participants) | 13 | 5 | 13 | 8 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 5 | 13 | 8 | 39
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.73 (1.44) | 9.48 (1.17) | 9.35 (1.41) | 9.28 (1.48) | 9.145 (1.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 13 | 5 | 13 | 8 | 39
Region of Enrollment [Number; unit: participants]
  United States | 13 | 5 | 13 | 8 | 39

OUTCOME MEASURES:

1. Primary Outcome: Beta-carotene Levels Between Overweight and Lean Boys at Baseline
Description: Value at baseline. Beta-carotene is a component of the body's natural defense system against every day oxidative stress. Beta-carotene concentrations were measured by reverse-phase high-performance liquid chromatography with photodiode array detection between 220-600 nm.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: mM/L
Groups:
- Overweight: Overweight boys prior to receiving intervention.
- Lean: Lean boys prior to receiving intervention.
Arm/Group | Overweight | Lean
Number analyzed (Participants) | 26 | 9
mM/L | 0.22 (0.16-0.36) [0.12 to 0.26] | 0.29 (0.12-0.26) [0.16 to 0.36]

2. Primary Outcome: Percent Change From Baseline in Beta-Carotene in Overweight and Lean Boys
Description: Value at 6 months minus value at baseline. Beta-carotene is a component of the body's natural defense system against every day oxidative stress. Beta-carotene concentrations were measured by reverse-phase high-performance liquid chromatography with photodiode array detection between 220-600 nm.
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Groups:
- Overweight FVJC: Results displayed for overweight boys who received 6 months of FVJC intervention
- Overweight Placebo: Reesults displayed for overweight boys who received 6 months of Placebo intervention
Arm/Group | Overweight FVJC | Lean FVJC | Overweight Placebo | Lean Placebo
Number analyzed (Participants) | 11 | 5 | 10 | 4
Percent Change | 334 (57) | 303 (85) | -30 (57) | 23 (94)

ADVERSE EVENTS:
Groups:
- Overweight FVJC: Overweight Boys receiving Fruit and Vegetable Juice Concentrate (FVJC), 1 capsule, twice a day, for 6 months.
- Lean FVJC: Lean Boys receiving Fruit and Vegetable Juice Concentrate (FVJC), 1 capsule, twice a day, for 6 months.
- Overweight Placebo: Overweight Boys receiving Placebo, 1 capsule, twice a day, for 6 months.
- Lean Placebo: Lean Boys receiving Placebo, 1 capsule, twice a day, for 6 months.
Arm/Group | Overweight FVJC | Lean FVJC | Overweight Placebo | Lean Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/5 | 0/13 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/5 | 0/13 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No